CLINICAL TRIAL: NCT02164435
Title: Effects of Renal Sympathetic Denervation on the Cardiac and Renal Functions in Patients With Drug-resistant Hypertension Through MRI Evaluation
Acronym: RDN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Adelaide (Other)
Responsible Party: Principal Investigator, Stephen Grant Worthley, Helpman Chair of Cardiovascular Medicine, University of Adelaide
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CI-12-044-AU-HT
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Uncontrolled Hypertension
Keywords: Uncontrolled hypertension; Renal denervation; Renal artery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Renal Denervation (Other)
  Interventions: Procedure: Renal Denervation (EnligHTN™) Renal artery ablation with the EnligHTN™ Renal Denervation System.

INTERVENTIONS:
Procedure: Renal Denervation (EnligHTN™) Renal artery ablation with the EnligHTN™ Renal Denervation System.

SUMMARY:
This is a prospective, single centre clinical investigation looking at short (6 months) and long term (24 months) changes in cardiac function and renal function in patients with drug-resistant hypertension post renal sympathetic denervation.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be able and willing to comply with the required follow-up schedule
* Therapeutic Goods Association approved indications for EnligHTN™ Renal Denervation System
* Subject is ≥ 18 years of age at time of consent Subject has office SBP ≥ 160 mmHg (except for subjects with Diabetes Mellitus who must demonstrate an office SBP of ≥ 150 mm Hg) within 14 days of the procedure ◦Subject is taking ≥ 3 antihypertensive medications concurrently at maximum tolerated dose (this must include one diuretic) or subject has a documented intolerance to at least 2 out of the 4 major classes of anti-hypertensives (ACE/ARB, CCB, Diuretics, Beta Blockers and is unable to take 3 antihypertensive drugs.

Exclusion Criteria:

* Standard CMR exclusions;

  * implanted cardiac device
  * intracranial metallic implants
  * claustrophobia -Gadolinium-specific: estimated GFR <60 mls/min (usual clinical cut-off is <30 mls/min).
* Adenosine-specific:

  * asthma / reactive airways disease
  * >first degree atrioventricular block
  * concomitant use of dipyridamole or theophylline consumption of caffeine within 48 hours of proposed investigation
  * EnligHTN™ Renal Denervation System exclusion criteria:

Subject has an identified cause of secondary hypertension

* Subject has an estimated GFR <45 mL/min per 1.73 m2 using the MDRD formula
* Subject has undergone prior renal angioplasty, indwelling renal stents, and/or aortic stent grafts
* Subject has haemodynamically significant valvular heart disease
* Subject has a life expectancy less than 12 months, as determined by the PI
* Subject is participating in another clinical study Subject is pregnant, nursing, or of childbearing potential and is not using adequate contraceptive methods
* Subject has renal arteries with diameter(s) < 4 mm in diameter

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-07 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Cardiac Function (evaluated by MRI) | Baseline and 6 Months
  MRI Indices of Cardiac Function
  * Myocardial mass and myocardial fibrosis
  * Atrial and ventricular ejection function
  * Myocardial perfusion
  * Arterial distensibility

SECONDARY OUTCOMES:
Renal Function (evaluated by MRI) | Baseline, 6 Months and 24 Months
  MRI Indices of Renal Function:
  * Renal blood flow
  * Renal perfusion
  * Urinary protein
Cardiac Function | Baseline and 24 Months
  MRI Indices of Cardiac Function
  * Myocardial mass and myocardial fibrosis
  * Atrial and ventricular ejection function
  * Myocardial perfusion
  * Arterial distensibility

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Adelaide Hospital Adelaide, Adelaide, South Australia, Australia

REFERENCES:
- [Derived] Delacroix S, Chokka RG, Nelson AJ, Wong DT, Pederson S, Nimmo J, Rajwani A, Williams K, Teo KS, Worthley SG. Effects of renal sympathetic denervation on myocardial structure, function and perfusion: A serial CMR study. Atherosclerosis. 2018 May;272:207-215. doi: 10.1016/j.atherosclerosis.2018.03.022. Epub 2018 Mar 10. PMID 29627741